CLINICAL TRIAL: NCT04916158
Title: Evaluation of the Effectiveness of an Accelerated Rehabilitation Protocol Based on Multimodal Analgesia Optimization for Uni-compartmental Knee Prosthesis Surgery: Observational, Prospective, Monocentric "Before-after"
Brief Title: Evaluation of the Effectiveness of an Accelerated Rehabilitation Protocol Based on Multimodal Analgesia Optimization for Uni-compartmental Knee Prosthesis Surgery
Acronym: APUC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0324
Record Dates: First submitted 2021-01-26; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia
Keywords: IPACK, knee arthroplasty, ambulatory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, prosthetic replacement for osteoarthritis of the knee is a frequent surgery. In France, nearly 100,000 knee arthroplasties are performed each year . Over the last two decades, there has been growing interest in performing single compartment knee replacement (SKR) surgery in patients with isolated single compartment osteoarthritis. The explanation lies in faster recovery, less postoperative pain and less morbidity compared to total knee arthroplasty (TKR) . Pain control is one of the major elements of outpatient management of CKD . Prosthetic knee surgery is very painful, the median pain is rated at 5 out of 10 and on average we use 32 milligrams of morphine . The efficiency of the adductor canal block is effective in this context, it avoids the motor block obtained by the femoral block, therefore interesting for ambulatory management in view of a resumption of the fast walking foreseen for the patient. The IPACK (interspace between popliteal artery and the capsule posterior knee) is designed to block the small sensory branches of the sciatic nerve that pass through this space without affecting the motor components. The IPACK block provides analgesia only for the posterior knee and would probably be ineffective alone for postoperative analgesia It is therefore often performed with an adductor canal block for multimodal analgesia. This block is performed in several facilities, and data are increasingly emerging on its effectiveness .

Thus, based on the recommendations of the French Society of Anesthesia and Resuscitation, on improved rehabilitation after heavy orthopedic surgery on the lower limb published in 2019 the objective of this study is to evaluate the relevance of a protocol concerning prosthetic knee replacement (PUC) in ambulatory care, based on optimized pain control.

DETAILED DESCRIPTION:
In France, nearly 100,000 knee arthroplasties are performed each year . Knee prostheses generate a functional benefit demonstrated in the literature and limited perioperative morbidity and mortality. Over the past two decades, there has been growing interest in the use of single-compartment knee arthroplasty (SKR) in patients with isolated single-compartment osteoarthritis (OA). The explanation lies in faster recovery, less postoperative pain and less morbidity compared to total knee arthroplasty (TKR) Improvements in perioperative care with regard to analgesia, anesthesia, but also nursing care and rehabilitation have led to a significant reduction in length of stay. Effective pain management is essential and is a necessary condition for early mobilization and a reduction in length of stay. Cross et al. and Berger et al. have shown that reducing the length of stay of patients hospitalized after knee arthroplasty can be achieved not only without compromising patient safety, but also without compromising patient satisfaction .

Anticipating pain control represents a major asset for ambulatory management. As early as the end of the 1990s, it was demonstrated that pain control is the main parameter in ambulatory surgery .prosthetic knee surgery is a very painful surgery. The efficiency of the adductor canal block is effective in this context. It reduces the motor block obtained at the level of the femoral block, which is particularly interesting for ambulatory management with a view to the patient's planned fast walking. The IPACK (interspace between popliteal artery and the capsule posterior knee) is designed to block the small sensory branches of the sciatic nerve that travel in this space without affecting the motor components. The IPACK block provides analgesia only for the posterior knee and would probably be ineffective alone for postoperative analgesia,so it is often performed with an adductor canal block in a multimodal analgesic pathway. Although this block is performed in several institutions, data is still emerging on its effectiveness. For example, a randomized trial in a single institution involving 86 patients undergoing GPT revealed that the combination of IPACK, adductor canal block and periarticular infiltration improved postoperative analgesia and reduced opioid consumption compared to periarticular injection alone .

Thus, based on the SFAR recommendations on improved rehabilitation after heavy orthopedic surgery on the lower limb published in 2019 , we set up a protocol for a feasibility study of prosthetic knee replacement (PUC) on an outpatient basis, based on optimized pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with programmed SKR,
* >18 and < 85 years of age,
* Score ASA 1-2,
* No cognitive impairment,
* No thromboembolic TCDA,
* Without CI to local anesthetics, analgesics,
* Accepting outpatient care
* No opposition formulated

Exclusion Criteria:

<18 years and >85 years

* Patients under legal protection (guardianship, curatorship, ...)
* Refusal to participate
* Support for a total knee prosthesis,
* Emergency surgery or revision surgery,
* ASA3-4,
* SAOS not fitted,
* Allergy or hypersensitivity to local anesthetics,
* Outpatient discharge criteria not met.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with programmed SKR
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Test get up and go test measured from day 0 to day 3. The test is successful if the score is >1 | Day 0 to Day 3

SECONDARY OUTCOMES:
evaluation of the patient's recovery by the QOR-15 questionnaire at 24 and 48 hours, | 24 and 48 hours
  quality of recovery
evaluation of visual analogue pain scale up to Day 5 postoperatively | day 5
evaluation of morphine consumption up to Day 5 postoperatively | day 5

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.